CLINICAL TRIAL: NCT02445963
Title: A Phase 1 Open-label, Dose Escalating Study of Artificial Shigella Flexneri 2a InvaplexAR Administered Intranasally to Healthy, Adult Volunteers to Evaluate Safety and Immunogenicity
Brief Title: Safety and Immunogenicity of Artificial Invaplex (Shigella Flexneri 2a InvaplexAR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-15-19; A-18716 (Other: Walter Reed Army Institute of Research); NMRC.2015.0003 (Other: Naval Medical Research Center)
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Shigellosis; Bacillary Dysentery
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 μg S. flexneri 2a Invaplex (Active Comparator): 10 subjects vaccinated on days 0, 14, 28
  Interventions: Biological: Shigella flexneri 2a InvaplexAR
- 50 μg S. flexneri 2a Invaplex (Active Comparator): 10 subjects vaccinated on days 0, 14, 28
  Interventions: Biological: Shigella flexneri 2a InvaplexAR
- 250 μg S. flexneri 2a Invaplex (Active Comparator): 10 subjects vaccinated on days 0, 14, 28
  Interventions: Biological: Shigella flexneri 2a InvaplexAR
- 500 μg S. flexneri 2a Invaplex (Active Comparator): 10 subjects vaccinated on days 0, 14, 28
  Interventions: Biological: Shigella flexneri 2a InvaplexAR

INTERVENTIONS:
Biological: Shigella flexneri 2a InvaplexAR — The investigational product is S. flexneri 2a InvaplexAR. The product is composed of three individual components IpaB, IpaC, and LPS. The components were assembled into the high molecular weight S. flexneri 2a InvaplexAR complex and subsequently purified by ion-exchange chromatography yielding a bulk lot.

SUMMARY:
This study is an open-label, dose-escalating Phase 1 investigation of S. flexneri 2a InvaplexAR vaccine. A total of up to 40 subjects will receive one of four S. flexneri 2a InvaplexAR vaccine doses. The vaccine will be administered intranasally (without adjuvant).

DETAILED DESCRIPTION:
The vaccine will be administered on Days 0,14, and 28. Volunteers (10 per group [8 minimum]) will receive the same dose at each vaccination dependent upon group assignment. Groups will be divided according to the table below. An interval no less than 1 week will separate the third dose of a group from the first dose of the next group (receiving an increased InvaplexAR dose). Blood, stool, and saliva specimens will be collected at pre-specified intervals to examine systemic and mucosal vaccine antigen-specific immune responses. Ocular tear samples will be collected in groups C and D. Vaccine safety will be actively monitored during vaccination and for 28 days following the third vaccine dose. The decision to advance to the next dose level is based on the safety assessment (not immunogenicity). A dose level with no occurrence of stopping criteria in the 7 days following the last vaccine dose will prompt moving to the next higher level. All safety data will be summarized and reviewed with the research monitor prior to dose escalation. In addition, a report of all safety data will be provided to the sponsor's safety office for informational purposes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved > 70% accuracy).
* Signed informed consent document.
* Available for the required follow-up period and scheduled clinic visits.
* Women: Negative pregnancy test with understanding (through informed consent process) to not become pregnant nor to breastfeed during the study or within 3 months following last vaccination

Exclusion Criteria:

* Health problems (for example, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension, or any other conditions that might place the subjects at increased risk of adverse events)- study clinicians, in consultation with the PI, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the Research Monitor as appropriate.
* Clinically significant abnormalities on physical examination (chronic sinusitis or seasonal rhinitis) which compromise identification and interpretation of potential vaccine associated adverse effects.
* Use of immunosuppressive and/or immunomodulative drugs such as corticosteroids or chemotherapeutics that may influence antibody development.
* Immunosuppressive illnesses (including IgA deficiency defined by serum IgA below level of detection or <7mg/dL).
* Participation in research involving another investigational product (defined as receipt of an investigational product or exposure to an invasive investigational device) 30 days before planned date of first vaccination or anytime throughout the duration of the study until the last study safety visit.
* Positive blood test for HBsAG, HCV, HIV-1/HIV-2.
* Clinically significant abnormalities on basic laboratory screening.
* Presence of significant unexplained laboratory abnormalities that in the opinion of the PI may potentially confound the analysis of the study results.
* Current smoker or smoker in past 1 year ('smoker' defined as daily cigarette, cigar, or pipe use for a period of at least 1 month).

Research specific

* Structural abnormalities on sinus/nasal cavity examination.
* Rhinoplasty.
* Nasal polyps.
* Nasal ulcers.
* Deviated nasal septum. This question is being used to determine whether the volunteer has a clinically significant deviated septum that causes nasal obstruction (thereby causing difficulty breathing), interferes with normal sinus drainage, or obscures visualization of the posterior nasal cavity complicating examination and safety monitoring..
* Chronic sinusitis/rhinitis.
* Current or planned use of nasal topical corticosteroids and/or nasal spray medications in the 4 weeks prior to dosing or during the study vaccination period.
* Current or recent history (in the past 5 years) of reactive airway disease (asthma), chronic obstructive pulmonary disease, or chronic bronchitis.
* History of Bell's palsy.
* Chronic use (weekly or more often) of anti-diarrheal, anti-constipation, or antacid therapy (excluding use associated with spicy meals).
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* Personal or family history of inflammatory arthritis.
* Positive blood test for HLA-B27.
* History of allergy to any vaccine.

Prior Exposure to Shigella

* Serum IgG titer ≥ 2500 to Shigella flexneri 2a LPS.
* History of microbiologically confirmed Shigella infection in the past 3 years.
* Received previous experimental Shigella vaccine or live Shigella challenge.
* Travel to countries with symptoms of travelers' diarrhea where Shigella or other enteric infections are endemic (most of the developing world) within the past 6 months prior to dosing.
* Occupation involving handling of Shigella bacteria currently, or in the past 3 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Duplessis, MD, MPH, MS, Principal Investigator — Enteric Diseases Department Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Clinical Trials Center, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Duplessis C, Clarkson KA, Ross Turbyfill K, Alcala AN, Gutierrez R, Riddle MS, Lee T, Paolino K, Weerts HP, Lynen A, Oaks EV, Porter CK, Kaminski R. GMP manufacture of Shigella flexneri 2a Artificial Invaplex (InvaplexAR) and evaluation in a Phase 1 Open-label, dose escalating study administered intranasally to healthy, adult volunteers. Vaccine. 2023 Oct 6;41(42):6261-6271. doi: 10.1016/j.vaccine.2023.08.051. Epub 2023 Sep 2. PMID 37666695

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 μg S. Flexneri 2a Invaplex; 50 μg S. Flexneri 2a Invaplex: 9 subjects vaccinated on days 0, 14, 28
  Shigella flexneri 2a InvaplexAR: The investigational product is S. flexneri 2a InvaplexAR. The product is composed of three individual components IpaB, IpaC, and LPS. The components were assembled into the high molecular weight S. flexneri 2a InvaplexAR complex and subsequently purified by ion-exchange chromatography yielding a bulk lot.
Period: Overall Study
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
Started | 9 | 9 | 10 | 10
Completed | 7 | 9 | 9 | 10
Not Completed | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Change in employment | 1 | 0 | 0 | 0
Not completed — Symptoms post-vaccination | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex | Total
Number analyzed (Participants) | 9 | 9 | 10 | 10 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [22 to 28] | 34 [26 to 42] | 28 [27 to 31] | 28 [24 to 36] | 28 [24 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 2 | 10
  Male | 7 | 4 | 9 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 8 | 9 | 10 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 4 | 9
  White | 7 | 6 | 9 | 6 | 28
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 10 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events
Description: Number of adverse events related to the vaccine for each arm
Time Frame: 166 days
Measure: Number; unit: Adverse Events
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
Number analyzed (Participants) | 9 | 9 | 10 | 10
Adverse Events | 27 | 37 | 41 | 46

2. Primary Outcome: Antibody Titers Against IgG and IgA Immunizing Antigens
Description: Serum samples will be assayed for antibody titers against the immunizing antigens LPS, IpaB, IpaC, and S. flexneri 2a Invaplex at screening, and Days 0, 14, 28, 35, 42, and 56 for 36 subjects. Previously established high-titer specimens will be included on each plate to track day to day interassay variation. For each antigen, pre- and post-vaccination serum samples will be assayed side-by-side. The antibody titer assigned to each sample will represent the geometric mean of duplicate tests performed on 2 different days. Reciprocal endpoint titers < 5 will be assigned a value of 2.5 for computational purposes. Seroconversion will be defined as a > 4-fold increase in endpoint titer between pre-and post-vaccination samples AND a post-vaccination reciprocal titer >10.
Time Frame: At screening and Days 0, 14, 28, 35, 42, and 56
Population: Subjects who received at least 2 vaccine doses were included in the immunology analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- 10 μg S. Flexneri 2a Invaplex: 8 subjects vaccinated on days 0, 14, 28
  Shigella flexneri 2a InvaplexAR: The investigational product is S. flexneri 2a InvaplexAR. The product is composed of three individual components IpaB, IpaC, and LPS. The components were assembled into the high molecular weight S. flexneri 2a InvaplexAR complex and subsequently purified by ion-exchange chromatography yielding a bulk lot.
- 250 μg S. Flexneri 2a Invaplex: 9 subjects vaccinated on days 0, 14, 28
  Shigella flexneri 2a InvaplexAR: The investigational product is S. flexneri 2a InvaplexAR. The product is composed of three individual components IpaB, IpaC, and LPS. The components were assembled into the high molecular weight S. flexneri 2a InvaplexAR complex and subsequently purified by ion-exchange chromatography yielding a bulk lot.
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
Number analyzed (Participants) | 8 | 9 | 9 | 10
titers
  Serum IgG (Invaplex) | 1345.4 [805.0 to 2248.8] | 4703.2 [2104.6 to 10510.2] | 5486.4 [2199.0 to 13688.0] | 5571.5 [2680.3 to 11581.5]
  Serum IgA (Invaplex) | 259.4 [108.4 to 620.7] | 800.0 [330.7 to 1935.6] | 685.8 [192.3 to 2445.5] | 606.3 [259.3 to 1417.4]
  Serum IgG (LPS) | 1902.7 [1138.4 to 3180.2] | 4703.2 [2434.3 to 9086.5] | 4703.2 [2939.8 to 7524.2] | 6400 [3056.1 to 13402.8]
  Serum IgA (LPS) | 259.4 [108.4 to 620.7] | 635.0 [330.6 to 1219.4] | 544.3 [207.5 to 1428.2] | 527.8 [233.3 to 1194.1]
  Serum IgG (IpaB) | 183.4 [103.3 to 325.7] | 740.7 [228.8 to 2397.8] | 342.9 [86.4 to 1361.0] | 229.7 [102.9 to 512.8]
  Serum IgA (IpaB) | 50.0 [NA to NA] — The data were not normally distributed | 73.5 [36.1 to 149.5] | 85.7 [42.8 to 171.5] | 50.0 [NA to NA] — The data were not normally distributed
  Serum IgG (IpaC) | 336.4 [171.2 to 660.7] | 2539.8 [1049.8 to 6145.1] | 1728.1 [353.8 to 8440.5] | 2599.2 [1049.6 to 6436.6]
  Serum IgA (IpaC) | 70.7 [38.1 to 131.4] | 317.5 [72.0 to 1399.2] | 272.2 [84.9 to 872.2] | 400.0 [144.4 to 1108.0]

3. Secondary Outcome: IgG and IgA Antigen-Specific Antibody Secreting Cell (ASC) Mucosal Responses
Description: ASC responses were assessed using isolated peripheral blood mononuclear cells (PBMCs). For each antigen, pre- and post-vaccination samples were tested on the same plates for total and vaccine-specific numbers. The ASC responses indirectly reflect intestinal immune responses through measurement of antigen-specific B-lymphocytes in systemic circulation before homing to gut effector sites. An ASC response was defined as > 10 ASCs above baseline.
Time Frame: 56 Days
Population: Arm 1: One patient was lost to follow-up post dose 1 vaccination, overall participants is therefore 8 for this arm Arm 3: One patient withdrew from the study due to symptoms post dose 1 vaccination, overall participants is therefore 9 for this arm
Measure: Median (95% Confidence Interval); unit: ASC per 10^6 PBMCs
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
Number analyzed (Participants) | 8 | 9 | 9 | 10
ASC per 10^6 PBMCs
  ASC IgG (Invaplex) | 0.5 [0.0 to 4.5] | 4.0 [3.0 to 9.0] | 5.0 [5.0 to 12.0] | 9.0 [4.0 to 17.0]
  ASC IgA (Invaplex) | 1.00 [1.0 to 2.0] | 27.0 [20.0 to 96.0] | 23.0 [15.0 to 62.0] | 41.5 [24.0 to 73.0]
  ASC IgG (LPS) | 0.0 [0.0 to 0.5] | 0.0 [0.0 to 0.0] | 1.0 [0.0 to 3.0] | 2.0 [0.0 to 9.0]
  ASC IgA (LPS) | 0.0 [0.0 to 0.0] | 4.0 [1.0 to 23.0] | 1.0 [0.0 to 7.0] | 3.0 [0.0 to 12.0]

4. Secondary Outcome: IgG and IgA Antigen-Specific Antibody Lymphocyte Supernatant (ALS) Mucosal Responses
Description: ALS responses were assessed using isolated peripheral blood mononuclear cells (PBMCs). For each antigen, pre- and post-vaccination samples were tested on the same plates for total and vaccine-specific numbers. The ALS responses indirectly reflect intestinal immune responses through measurement of antigen-specific B-lymphocytes in systemic circulation before homing to gut effector sites. An ALS response was defined as a ≥ 4-fold increase over baseline ALS titers.
Time Frame: 56 Days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
Number analyzed (Participants) | 8 | 9 | 9 | 10
fold change
  ALS IgG (Invaplex) | 1.2 [0.8 to 1.8] | 8.6 [2.5 to 29.7] | 9.3 [2.9 to 30.5] | 7.0 [2.8 to 17.6]
  ALS IgA (Invaplex) | 1.3 [0.7 to 2.4] | 8.6 [2.4 to 30.5] | 3.7 [1.3 to 10.9] | 4.3 [1.7 to 10.7]
  ALS IgG (LPS) | 1.2 [0.8 to 1.8] | 2.9 [1.4 to 6.0] | 4.0 [1.9 to 8.5] | 3.5 [1.8 to 6.7]
  ALS IgA (LPS) | 1.1 [0.9 to 1.3] | 3.2 [1.5 to 6.7] | 2.0 [1.2 to 3.4] | 2.1 [1.2 to 3.9]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 8 months
Description: Vaccine-related (possibly, probably, definitely) surveyed signs and symptoms of all study subjects receiving at least one dose of investigational product was assessed through targeted physical exams, symptom surveys, and other adverse events (AE) monitoring. Subjects were observed in clinic for 30 minutes, 24 hours, and 7days post vaccination to review their symptom diaries and to report any AEs. All vaccine-related and unrelated (not related, unlikely) AEs were reported.
Arm/Group | 10 μg S. Flexneri 2a Invaplex | 50 μg S. Flexneri 2a Invaplex | 250 μg S. Flexneri 2a Invaplex | 500 μg S. Flexneri 2a Invaplex
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 μg S. Flexneri 2a Invaplex (N=9) | 50 μg S. Flexneri 2a Invaplex (N=9) | 250 μg S. Flexneri 2a Invaplex (N=10) | 500 μg S. Flexneri 2a Invaplex (N=10)
AST Elevation (Investigations) | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 4 | 3
Fatigue (General disorders) | 3 | 2 | 2 | 4
Fever (General disorders) | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 4 | 5
Itchy Eyes (Eye disorders) | 0 | 2 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Nasal Burning (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 6 | 10
Nasal Itching (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 2
Nasal Mucosal Hyperemia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 6 | 2
Nasal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Stuffiness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal Tenderness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 4
Pharyngitis (Infections and infestations) | 3 | 1 | 4 | 7
Post-Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 9
Pulmonary Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 7 | 6
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 5
Tearing Eyes (Eye disorders) | 0 | 1 | 0 | 0
Upper Respiratory Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Abdominal Cramps (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2
BUN Elevation (Investigations) | 0 | 0 | 0 | 1
Chest Tightness (Unknown Etiology) (General disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dry Chapped Lips (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hemoglobinemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Joint Aches (Left Knee and Left Elbow) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lightheadedness (Nervous system disorders) | 1 | 0 | 0 | 0
Loose Stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Low Hemoglobin (Investigations) | 0 | 0 | 1 | 0
Lymphocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Olecranon bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Right Hip Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Right Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Right Upper Lip Fever Blister (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Systolic Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Urinary Tract Infection (UTI) (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No